CLINICAL TRIAL: NCT00590200
Title: Molecular Determinants of Coronary Artery Disease
Brief Title: GeneBank at the Cleveland Clinic: Molecular Determinants of Coronary Artery Disease
Acronym: GATC
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Millennium Pharmaceuticals, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stanley L Hazen, MD, PhD, Section Head, Preventive Cardiology & Rehabilitation; Chair, Department of Cardiovascular and Metabolic Sciences; Director, Center for Microbiome & Human Health, The Cleveland Clinic
Other Study IDs: IRB 4265; 5P50HL077107-02 (NIH); IRB 4265 (Other: Institutional Review Board); GeneBank (Other: Cleveland Clinic Foundation)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
Keywords: CAD; Cardiovascular Disease; CVD; MI; Myocardial Infarction; Heart Attack; CABG; Revascularization; genetic
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 70 mls of blood will be dispensed as follows (Approximately 80 mls if cell lines are drawn or if the patient is having a cardiac CT scan):
  4 x 10 mls EDTA Tube (DNA will be amplified in order to preserve quantity)
  1. x 10ml Lithium Heparin Tube (drawn on selected patient populations at CCF only- See Appendix E. for cell line protocol)
  2. x 5 mls Serum Tube
  1 x 7 mls Serum Tube
  1 x 2.7 mls Sodium Citrate Tube (CCF Only. See Appendix D)
  1 x 4.5 mls CTAD tube (platelet release inhibited)
  1 x 4.5 mls SCAT-1 tube (coagulation activation inhibited) (Blood may be dispensed in the above tubes in different quantities if functional studies are needed on a subset of samples)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This proposal delineates a research plan to collect blood from patients undergoing heart catheterization or who have had a heart catheterization within one year and are coming in for outpatient appointments, or who have scheduled cardiac CT scans at the Cleveland Clinic over a five-year period for the purpose of establishing a gene bank registry. In addition, the University of North Carolina at Chapel Hill will enroll 1,000 non-Caucasian patients and MetroHealth Medical center in Cleveland will enroll 1,000 non-Caucasian patients. The blood collected will be processed to create a repository of DNA, lymphoblastoid cell line immortalization on selected patient populations, plasma and serum. The DNA will be amplified in certain patient populations to preserve the quantity. Along with a sample of blood collected from individual patients, a concise general medical history, demographic data, electrocardiographic data, echocardiographic data (available for about 55% of patients at the present time), and laboratory data will be collected. A short interview will take place after enrollment during the outpatient visit or hospital stay, or may be conducted via phone call after enrollment. All the clinical data gathered will be compiled in GATC heart center database, and would be stored in a format where a culmination of clinical findings, i.e. representing a disease of interest, can be used to search the database to identify the blood samples of all patients with such characteristics for further study.

DETAILED DESCRIPTION:
The study is to commence on March 1st 2001 and is to be completed within 2-5 years. The targeted number of patients to be enrolled is 15,000. All patients undergoing cardiac catheterization or have had a heart catheterization within one year, coming in for outpatient appointments, or have scheduled cardiac CT scans or CT scans performed within one year of scheduled blood draw, will be eligible to be enrolled. Patients inclusion criteria are as follows, once informed consent is obtained:

1. Males or females at least 18 years old.
2. Patient has not been previously enrolled in the genebank registry.
3. Patient able to give informed consent.
4. Patient to undergo cardiac catheterization or had a left heart cath at The Cleveland Clinic or at The University of North Carolina at Chapel Hill, or at MetroHealth Medical Center within 1 year.
5. Patients > or = to 50 y/o with normal cardiac catheterizations (< 30% in all coronary vessels per angio). (If subjects enrolled as normal controls are later deemed to have significant Coronary Artery Disease (CAD), the subject's blood and data will still be useful in the GeneBank under the broader scope of the study)
6. Any patient with history of myocardial infarction (MI). (If a subject reports history of MI at another facility, outside records will be obtained to confirm the diagnosis. If MI cannot be confirmed by data in the record, the subject's blood and data will still be useful in the Genebank under the broader scope of the study.)
7. Non-Caucasian patients or of Hispanic Ethnicity (UNC and MetroHealth Medical Center only)
8. All Patients undergoing Cardiac CT or had Cardiac CT within 1 year (CCF only)
9. Any patient coming to the Heart and Vascular Institute for outpatient scheduled appointments.
10. Any patients that have had or are going to have an implanted cardioverter defibrillator (ICD) or cardiac resynchronization defibrillator (CRT-D).
11. Any patients with cardiac arrhythmias or a family history of cardiac arrhythmias.

(Cleveland Clinic will follow inclusion criteria 1-6 and 8-11, UNC and MetroHealth Medical Center will follow criteria 1-11).

Exclusion criteria:

None except as in Inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years old.
2. Patient has not been previously enrolled in the genebank registry.
3. Patient able to give informed consent.
4. Patient to undergo cardiac catheterization or had a left heart cath at The Cleveland Clinic or at The University of North Carolina at Chapel Hill, or at MetroHealth Medical Center within 1 year.
5. Patients > or = to 50 y/o with normal cardiac catheterizations (< 30% in all coronary vessels per angio). (If subjects enrolled as normal controls are later deemed to have significant CAD, the subject's blood and data will still be useful in the Genebank under the broader scope of the study).
6. Any patient with history of myocardial infarction. (If a subject reports history of MI at another facility, outside records will be obtained to confirm the diagnosis. If MI cannot be confirmed by data in the record, the subject's blood and data will still be useful in the Genebank under the broader scope of the study).
7. Non-caucasian patients or of Hispanic Ethnicity (UNC and MetroHealth Medical; Center only).
8. All Patients undergoing Cardiac CT or had Cardiac CT within 1 year (CCF only). (Cleveland Clinic will follow inclusion criteria 1-7, 9, UNC and MetroHealth Medical Center will follow criteria1-8).
9. Any patients coming to the Heart and Vascular Institute for outpatient scheduled appointments.
10. Any patients that have had or are going to have an implanted cardioverter defibrillator (ICD) or Cardiac Resynchronization Defibrillator (CRT-D).
11. Any patients with cardiac arrhythmias or a family history of cardiac arrhythmias.

Exclusion Criteria:

None except as noted in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Cleveland Clinic patients undergoing cardiac catheterization or have had a heart catheterization within one year, coming in for outpatient appointments, or have scheduled cardiac CT scans or CT scans performed within one year of scheduled blood draw, will be eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 9880 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2007-07 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Coronary Artery Disease | 3 years
  Development of Coronary Artery Disease

SECONDARY OUTCOMES:
Death | 5 years
  All cause mortality
Revascularization | 3 years
  Need for revascularization
Percutaneous Coronary Intervention/Stent | 3 years
  Need for percutaneous coronary intervention and/or stent
Myocardial Infarction | 3 years
  New myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hazen, MD, PhD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witkowski M, Wu Y, Hazen SL, Tang WHW. Prognostic value of subclinical myocardial necrosis using high-sensitivity cardiac troponin T in patients with prediabetes. Cardiovasc Diabetol. 2021 Aug 21;20(1):171. doi: 10.1186/s12933-021-01365-9. PMID 34419046
- [Derived] Dupont M, Wu Y, Hazen SL, Tang WH. Cystatin C identifies patients with stable chronic heart failure at increased risk for adverse cardiovascular events. Circ Heart Fail. 2012 Sep 1;5(5):602-9. doi: 10.1161/CIRCHEARTFAILURE.112.966960. Epub 2012 Aug 16. PMID 22899766